CLINICAL TRIAL: NCT02741453
Title: Scanning of Bilateral Internal Jugular Veins With Ultrasound Prior to CVC Placement - Effect on Success and Complications
Brief Title: Bilateral Internal Jugular Veins Ultrasound Scanning Prior to CVC Placement
Acronym: BIUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Ryan Story, Resident, Vanderbilt University Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 160704
Record Dates: First submitted 2016-04-14; First posted 2016-04-18 (Estimated); Last update posted 2017-07-14 (Actual); Status verified 2017-07

CONDITIONS: Central Venous Catheterization; Ultrasonography; Critical Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Practice (Active Comparator): Placement of a CVC by standard practice
  Interventions: Procedure: Standard Practice
- Bilateral IJ Ultrasound Scanning (Experimental): Placement of a CVC after mandatory ultrasound scanning of both right and left internal jugular veins
  Interventions: Procedure: Bilateral IJ Ultrasound Scanning

INTERVENTIONS:
Procedure: Standard Practice
  Arms: Standard Practice
Procedure: Bilateral IJ Ultrasound Scanning
  Arms: Bilateral IJ Ultrasound Scanning

SUMMARY:
Central venous catheter placement is a common procedure in the intensive care unit and is a required skill for all residents working in the critical care setting. Central venous catheters (CVC) are placed for a variety of reasons including administration of caustic medications, administration of fluids or blood products for rapid resuscitation, access for hemodynamic monitoring or transvenous pacing, temporary vascular access for dialysis, or inability to obtain peripheral IV access. CVC's are routinely placed in the internal jugular vein in the Vanderbilt medical ICU and ultrasound guidance is used. Placement of the CVC on the right IJ instead of the left IJ is commonly preferred due to the more direct path to the superior vena cava. However, placement in the left IJ may be necessary for a variety of reasons. The investigators intend to compare the standard practice of residents and nurse practitioners placing IJ CVCs in the medical ICU against mandatory screening of the right and left IJ prior to selection of the CVC placement site. The investigators will accomplish this by assessing the relative first pass stick and overall success rates, the rate of aborted procedures, and the rate of complications between standard practice and mandatory screening of bilateral internal jugular veins prior to CVC site selection.

DETAILED DESCRIPTION:
Central venous catheter placement is a common procedure in the intensive care unit and is a required skill for all residents working in the critical care setting. Central venous catheters (CVC) are placed for a variety of reasons including administration of caustic medications, administration of fluids or blood products for rapid resuscitation, access for hemodynamic monitoring or transvenous pacing, temporary vascular access for dialysis, or inability to obtain peripheral IV access.

The 2011 CDC Guidelines for Prevention of Intravascular Catheter-Related Infections recommends placement of a CVC in the subclavian vein rather than the internal jugular vein to minimize infection risk. However, due to lack of experience with placement in the subclavian vein, in the Vanderbilt MICU, it is most common for residents to place catheters in the internal jugular vein. Placement of the CVC under ultrasound guidance has become standard of care and is also recommended by the aforementioned CDC guidelines (CDC guidelines).

Ultrasound guidance for CVC placement has improved patient safety by reducing the rate of complications, improving success rates, and decreasing number of attempts and time for successful insertion (Brass). The benefit of ultrasound guidance in reducing complications is especially important when less experienced operators such as residents are placing a CVC (Rando, Airapetian, Dodge). The addition of an ultrasound machine to an otherwise sterile procedure does not increase the rate of catheter associated blood stream infections (Cartier).

Placement of the IJ CVC on the right instead of the left is commonly preferred due to the more direct path to the superior vena cava. However, placement in the left IJ may be necessary for a variety of reasons. Depending on head position, the degree of overlap between the right IJ and the right carotid artery may make right sided placement precarious due to risk of arterial puncture (Ozbek, Maecken). Previously undetected IJ thrombus on the right may also prevent CVC placement, requiring a switch to the contralateral side (Goel). Ultrasound guidance could also reveal a unilateral vascular anatomic anomaly that would otherwise complicate CVC insertion (Benter, Rossi).

For these reasons, the investigators intend to compare the standard practice of residents placing IJ CVC in the medical ICU against mandatory screening of the right and left IJ prior to selection of the CVC placement site.

The benefits of ultrasound guidance for IJ CVC placement are well established. However, the benefits of ultrasound guidance may be extended by more fully evaluating both the left and right IJ prior to choosing a side for placement. As mentioned previously, several factors could make placement of the CVC on a particular side either more successful or precarious. These factors include possible asymmetric diameter of the IJ vein, unfavorable relationship of the IJ to the carotid artery, pre-existing IJ thrombus, or other aberrant vascular anatomy.

This study will begin with a 4 month period of data collection on the standard practice of IJ CVC placement by residents in the medical intensive care unit. Data will be collected on the success rate of CVC insertion as measured by "first stick" placement of the catheter. The study will also record how often placement of the CVC must be aborted in favor of an attempt on the contralateral side. Any incidental detection of pre-existing conditions that could complicate CVC placement, including IJ thrombus or aberrant anatomy, will also be recorded. Finally, the investigators will record rates of immediate complication of CVC placement, including pneumothorax, hemothorax, and arterial placement or puncture of the CVC catheter.

In the medical ICU of the institution where this study will occur, nurse practitioners perform similar duties to residents on a separate but similarly operating ICU team. Data on central line placement by nurse practitioners will also be collected.

The specific aims will be threefold:

Specific Aim 1: To assess the first pass and overall success rates when both IJ veins are evaluated by ultrasound compared to standard IJ CVC placement by ultrasound.

Specific Aim 2: To assess the rate of aborted procedures between the two study periods, as defined by failure of catheter placement at the side of first needle puncture site or failure of catheter placement overall.

Specific Aim 3: To assess the rate of complications when IJ central venous catheters are placed after evaluation of bilateral IJ sites compared to current practice of placing IJ catheters under ultrasound guidance.

ELIGIBILITY:
Inclusion Criteria:

* Patient admitted to the medical intensive care unit on the 8th floor
* Central venous catheter placed by a resident or nurse practitioner working in the medical intensive care unit
* Central venous catheter placed in the right or left internal jugular vein
* Central venous catheter placed with ultrasound guidance

Exclusion Criteria:

* Line placed outside the MICU
* Placed in the subclavian or femoral vein
* Placed by a fellow in training or attending physician
* Placed under emergent or time-sensitive conditions
* Placed during a code
* Placed under non-sterile conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 278 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2017-05-01 (Actual); Study Completion 2017-05-01 (Actual)

PRIMARY OUTCOMES:
First Pass Success Rate | 8 months
  First pass success rate will be defined as access of the initially targeted internal jugular vein with the first pass of the guide needle.

SECONDARY OUTCOMES:
Success Rate | 8 months
  Success rate will be defined as successful placement of the central venous catheter at the initially targeted site.
Aborted Procedure Rate | 8 months
  Aborted procedure will be defined as failure to place the catheter at side of first needle puncture site or failure of catheter placement overall.
Complication Rate | 8 months
  Complications will include but will not be confined to the following:
  * Catheter related infection
  * Catheter related thrombosis
  * Injury to adjacent vascular structures
  * Arterial placement of central venous catheter
  * Arrhythmia induced by catheter placement
  * Violation of the pleural space resulting in pneumothorax or hemothorax
  * Venous air embolism
  * Uncontrolled bleeding from placement including bleeding compromising the airway

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Story, MD, Principal Investigator — Vanderbilt University Medical Center; Todd Rice, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] O'Grady NP, Alexander M, Burns LA, Dellinger EP, Garland J, Heard SO, Lipsett PA, Masur H, Mermel LA, Pearson ML, Raad II, Randolph AG, Rupp ME, Saint S; Healthcare Infection Control Practices Advisory Committee. Guidelines for the prevention of intravascular catheter-related infections. Am J Infect Control. 2011 May;39(4 Suppl 1):S1-34. doi: 10.1016/j.ajic.2011.01.003. No abstract available. PMID 21511081
- [Background] Brass P, Hellmich M, Kolodziej L, Schick G, Smith AF. Ultrasound guidance versus anatomical landmarks for subclavian or femoral vein catheterization. Cochrane Database Syst Rev. 2015 Jan 9;1(1):CD011447. doi: 10.1002/14651858.CD011447. PMID 25575245
- [Background] Rando K, Castelli J, Pratt JP, Scavino M, Rey G, Rocca ME, Zunini G. Ultrasound-guided internal jugular vein catheterization: a randomized controlled trial. Heart Lung Vessel. 2014;6(1):13-23. PMID 24800194
- [Background] Airapetian N, Maizel J, Langelle F, Modeliar SS, Karakitsos D, Dupont H, Slama M. Ultrasound-guided central venous cannulation is superior to quick-look ultrasound and landmark methods among inexperienced operators: a prospective randomized study. Intensive Care Med. 2013 Nov;39(11):1938-44. doi: 10.1007/s00134-013-3072-z. Epub 2013 Sep 12. PMID 24026296
- [Background] Dodge KL, Lynch CA, Moore CL, Biroscak BJ, Evans LV. Use of ultrasound guidance improves central venous catheter insertion success rates among junior residents. J Ultrasound Med. 2012 Oct;31(10):1519-26. doi: 10.7863/jum.2012.31.10.1519. PMID 23011614
- [Background] Cartier V, Haenny A, Inan C, Walder B, Zingg W. No association between ultrasound-guided insertion of central venous catheters and bloodstream infection: a prospective observational study. J Hosp Infect. 2014 Jun;87(2):103-8. doi: 10.1016/j.jhin.2014.03.009. Epub 2014 Apr 13. PMID 24811115
- [Background] Ozbek S, Apiliogullari S, Kivrak AS, Kara I, Saltali AO. Relationship between the right internal jugular vein and carotid artery at ipsilateral head rotation. Ren Fail. 2013;35(5):761-5. doi: 10.3109/0886022X.2013.789970. Epub 2013 May 7. PMID 23650892
- [Background] Maecken T, Marcon C, Bomas S, Zenz M, Grau T. Relationship of the internal jugular vein to the common carotid artery: implications for ultrasound-guided vascular access. Eur J Anaesthesiol. 2011 May;28(5):351-5. doi: 10.1097/EJA.0b013e328341a492. PMID 21150630
- [Background] Goel S, Majhi S, Panigrahi B. Unexpected detection of internal jugular vein thrombus during ultrasound-guided central venous cannulation. J Cardiothorac Vasc Anesth. 2011 Oct;25(5):e36-7. doi: 10.1053/j.jvca.2011.03.177. Epub 2011 Jun 8. No abstract available. PMID 21641820
- [Background] Benter T, Teichgraber UK, Kluhs L, Papadopoulos S, Kohne CH, Felix R, Dorken B. Anatomical variations in the internal jugular veins of cancer patients affecting central venous access. Anatomical variation of the internal jugular vein. Ultraschall Med. 2001 Feb;22(1):23-6. doi: 10.1055/s-2001-11243. PMID 11253552
- [Background] Rossi UG, Rigamonti P, Torcia P, Mauri G, Brunini F, Rossi M, Gallieni M, Cariati M. Congenital anomalies of superior vena cava and their implications in central venous catheterization. J Vasc Access. 2015 Jul-Aug;16(4):265-8. doi: 10.5301/jva.5000371. Epub 2015 Mar 9. PMID 25768048